CLINICAL TRIAL: NCT06813963
Title: A Randomized, Double-Blind, Multicenter, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Minoxidil in the Repigmentation of White Hair in Adults
Brief Title: Minoxidil for Treating White Hair: A Randomized Controlled Trial
Acronym: MTWH-RCT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Wangzehao He, Doctoral Student in Plastic Surgery, Southern Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Minoxidil treats white hair
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-02

CONDITIONS: Grey Hair
Keywords: white hair

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5%minoxidil group (Experimental): Participants will apply high concentration Minoxidil (e.g., 5% Minoxidil solution) to the scalp twice daily for 12 months. The main purpose of the treatment is to evaluate the efficacy of high-concentration Minoxidil for treating non-pathological graying and to monitor its safety and tolerability.
  Interventions: Drug: Topical Minoxidil（5%） to the scalp.
- Placebo Group (Placebo Comparator): This group will receive a placebo solution (similar in appearance and odor to Minoxidil but without the active ingredient), applied to the scalp twice daily for 12months. This placebo group will serve as a control for comparing the effects of Minoxidil on non-pathological graying of hair.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topical Minoxidil（5%） to the scalp. — The patient will apply 5% Minoxidil topical solution to the scalp twice daily, with 7 sprays (approximately 1 mL) per application, for a duration of 12 months.
  Arms: 5%minoxidil group
Drug: Placebo — The patient will apply placebo to the scalp twice daily, with 7 sprays (approximately 1 mL) per application, for a duration of 12 months.
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to evaluate whether topical Minoxidil can restore hair pigmentation in individuals with non-pathological graying hair. The study population includes male and female participants aged [18to65] who have non-pathological graying of hair, meaning their graying is not due to any underlying medical conditions.

The main questions it aims to answer are:

Does topical Minoxidil improve hair pigmentation in individuals with non-pathological graying hair? What medical problems do participants have when topical use minoxidil? Researchers will compare participants receiving topical Minoxidil to those receiving a placebo to determine whether Minoxidil has a significant effect on restoring hair pigmentation.

Participants will:

Topical use minoxidil or a placebo twice a day for 12 months Visit the clinic once every months for checkups and tests Report any adverse effects or changes in hair characteristics throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The patients included in the study were those with a visible gray hair grading score of 2 or higher at screening and baseline visits, with depigmented hair shafts observable under dermoscopy.

Exclusion Criteria:

* Exclusion criteria included various pathological types of gray hair (including, but not limited to, alopecia areata, albinism, radiation-induced gray hair, and vitiligo); any scalp skin diseases (including, but not limited to, androgenetic alopecia, folliculitis, seborrheic dermatitis, psoriasis, tinea capitis, and scalp sebaceous cysts); and any history of medication use or other treatments applied to the scalp within the past year (including, but not limited to, minoxidil, hair transplantation surgery, boric acid lotion, ketoconazole shampoo, and corticosteroid ointments). Patients with severe systemic diseases, immune diseases, endocrine disorders, or neurological diseases were also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Reduction in the appearance gray hair grade | From enrollment to the end of treatment at 12 months
  we divided gray hair appearance into 11 progressive levels of severity, ranging from grade 0: fully pigmented, to grade 10: completely unpigmented.Two trained physicians (blinded to the trial group assignments) used a gray hair appearance color scale to rate patients' gray hair appearance to determine whether the primary outcome definition was met.

SECONDARY OUTCOMES:
Reduction 2 level in the appearance gray hair grade | From enrollment to the end of treatment at 12 months
  We divided gray hair appearance into 11 progressive levels of severity, ranging from grade 0: fully pigmented, to grade 10: completely unpigmented.Two trained physicians (blinded to the trial group assignments) used a gray hair appearance color scale to rate patients' gray hair appearance to determine whether the primary outcome definition was met.
White hair percent change from baseline | From enrollment to the end of treatment at 12 months
  We used tattoo to mark the patient's scalp and temporal areas, and observed the number of gray and black hairs at the marked locations using a dermatoscope. During each follow-up, we reassessed the gray-to-black hair ratio and any changes in hair pigmentation at the marked areas
Grayscale change | From enrollment to the end of treatment at 12 months
  During each follow-up, we photographed the patient's appearance and used ImageJ software to measure the grayscale value of the hair in the patient's appearance photos.
Amount of repigment white hair | From enrollment to the end of treatment at 12 months
  During each follow-up, we photographed the patient's appearance and used ImageJ software to measure the grayscale value of the hair in the patient's appearance photos.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First People's Hospital of Zhaoqing, Zhaoqing, Guangdong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP